CLINICAL TRIAL: NCT00080080
Title: Phase 2 Study of Talabostat and Docetaxel in Advanced Non-Small Cell Lung Cancer
Brief Title: Study of Talabostat and Docetaxel in Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Point Therapeutics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTH-302
Record Dates: First submitted 2004-03-23; First posted 2004-03-24 (Estimated); Last update posted 2007-06-08 (Estimated); Status verified 2007-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — talabostat; Tablets; Docetaxel

INTERVENTIONS:
Drug: talabostat (PT-100) tablets
Drug: Docetaxel

SUMMARY:
The purpose of this study is to determine the antitumor activity (response rate, time to tumor progression, survival) and safety of docetaxel in combination with talabostat in patients with advanced non-small cell lung cancer (NSCLC) who have failed a prior platinum-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Stage IIIb/IV NSCLC
* Failed or relapsed after receiving a platinum-containing chemotherapy regimen as first-line therapy for advanced NSCLC
* Measurable disease
* ECOG Performance Status of 0 or 1
* Expected survival ≥12 weeks
* Provide written informed consent

Exclusion Criteria:

* More than 2 prior chemotherapy regimens
* Brain metastases (exception: patients who have had a resection and/or completed a course of cranial irradiation, have no worsening CNS symptoms, and have discontinued all corticosteroids for that indication for at least 1 month)
* Any malignancy within the 5 years immediately prior to the first dose of study medication with the exception of basal cell or non-metastatic squamous cell carcinoma of the skin, and carcinoma in-situ of the cervix
* The need for chronic (i.e., >7 days) oral or intravenous corticosteroid therapy
* A history of severe hypersensitivity reactions to drugs formulated with polysorbate 80
* A history of myocardial infarction within 1 year of study entry, CABG within 6 months of study entry, severe congestive heart failure (ejection fraction <30%), history of ventricular arrhythmia, or other uncontrolled cardiac arrhythmia
* Any comorbidity or condition which, in the opinion of the investigator, may interfere with the assessments and procedures of this protocol
* Patients who are within 30 days of chemotherapy, radiation therapy, immunotherapy, or other investigational medication for NSCLC. Patients must have recovered from all of the side effects of treatment in order to be enrolled.
* Pregnant or lactating women.
* Clinically significant laboratory abnormalities, specifically:

Total bilirubin ≥institutional upper limit of normal (ULN); Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥1.5 x ULN concomitant with alkaline phosphatase >2.5 x ULN; Hepatitis B surface antigen or antibody to Hepatitis C (anti-HCV antibody); Serum creatinine ≥2.0mg/dL; or Granulocytes <1500/μL or platelets <100,000/μL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Cancer Center of Florida, Ocoee, Florida
  - University of Chicago, Chicago, Illinois
  - Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - New York Oncology/Hematology--Albany Regional Cancer Center, Albany, New York
  - Mt. Sinai School of Medicine, New York, New York
  - USB Cancer Center-- Nyack Hospital, Nyack, New York
  - Dayton Oncology & Hematology, Kettering, Ohio
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Cancer Care Northwest, Spokane, Washington